CLINICAL TRIAL: NCT06350422
Title: Neuroimage Genome Study of Neuroplasticity Associated With Microgravity
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Director and Clinical Professor, Chinese PLA General Hospital
Other Study IDs: Microgravity-ChinaPLAGH
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Microgravity; Neuroplasticity; MRI; Repeatable Battery for the Assessment of Neuropsychological Status
Keywords: Microgravity; Neuroplasticity; MRI; Repeatable Battery for the Assessment of Neuropsychological Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Head-Down tilt Bed Rest test — All of the volunteers underwent 60 days of the Head-Down tilt Bed Rest test.

SUMMARY:
This clinical trial investigates the neuroplasticity and cognitive status changes of the human brain in microgravity. To explore the relationship between cognitive status changes and brain functional activities, gray matter and white matter changes under microgravity exposure, screen and identify representative image markers, so as to provide decision-making information for the cognitive status changes of relevant personnel under microgravity environment.

DETAILED DESCRIPTION:
MRI has the advantage of non-invasive and non-radiation, and imaging the human brain after exposure to microgravity can reveal the neuroplastic changes in the astronaut's brain and discover the characteristics of functional activities behind it. The purpose of this study is to explore the image features and cognitive state related information related to the changes of human brain neuroplasticity under microgravity environment, and to identify the related image markers. At the same time, the pathophysiological mechanism is preliminarily discussed in this study. This study is helpful for us to explore the sensitivity of different brain structures and brain functions to space microgravity environment, so as to further understand the role and influence of space missions on brain health.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18-60 years
* No mental or other neurological disorders, no history of drug or alcohol abuse
* Generally in good condition, no clear major physical diseases, no hearing disorders
* No metal foreign bodies in the body, no contraindications to MRI scanning
* No claustrophobia
* Agree to participate in the clinical study and sign the informed consent

Exclusion Criteria:

* There are electronic implants or metal foreign bodies, such as cardiac pacemakers
* People with aneurysm surgery and intracranial aneurysm clip
* People who have had heart surgery and used artificial heart valves
* Having family planning
* Uncontrolled epilepsy or mental illness, can't cooperate with MRI examination
* Severe claustrophobia, can't cooperate with magnetic resonance examination
* Other circumstances that the clinical trial personnel consider inappropriate to participate in the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers who underwent 60 days of the Head-Down tilt Bed Rest test.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Local brain functional activity | 60 days after the Head-Down tilt Bed Rest test
  Based on resting-state functional MRI images, the changes of local brain functional activity before and after the Head-Down tilt Bed Rest test were compared.
Brain functional connectivity | 60 days after the Head-Down tilt Bed Rest test
  Based on resting-state functional MRI images, the changes of brain functional connectivity before and after the Head-Down tilt Bed Rest test were compared.
Brain structure - Morphology | 60 days after the Head-Down tilt Bed Rest test
  Based on 3D-T1WI, the changes of brain structure before and after the Head-Down tilt Bed Rest test were compared.
Brain fiber bundle and brain Diffusion index | 60 days after the Head-Down tilt Bed Rest test
  Based on diffusion tensor imaging, the changes of brain fiber bundle and brain diffusion index before and after the Head-Down tilt Bed Rest test were compared.
Brain blood flow | 60 days after the Head-Down tilt Bed Rest test
  Based on arterial spin labeling, the changes of brain blood flow before and after the Head-Down tilt Bed Rest test were compared.
Imaging indexes and clinical scale scores | 60 days after the Head-Down tilt Bed Rest test
  Based on the changes of relevant imaging indexes and the changes of relevant clinical scale scores, explore the correlation between the changes of relevant imaging indexes and relevant clinical scales scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China